CLINICAL TRIAL: NCT03693131
Title: MND-2119 Phase 3 Study to Evaluate the Efficacy and Safety of MND-2119 Compared to EPADEL CAPSULES 300 in Patients With Hypertriglyceridemia
Brief Title: Efficacy of MND-2119 in Participants With Hypertriglyceridemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mochida Pharmaceutical Company, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MND2119H31; JapicCTI-184130 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2018-09-30; First posted 2018-10-02 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia | interventions — Eicosapentaenoic Acid; eicosapentaenoic acid ethyl ester

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MND-2119 2 g (Experimental): MND-2119 2 g, orally, once daily after breakfast for 12 weeks.
  Interventions: Drug: Icosapent (MND-2119)
- MND-2119 4 g (Experimental): MND-2119 4 g, orally, once daily after breakfast for 12 weeks.
  Interventions: Drug: Icosapent (MND-2119)
- EPADEL CAPSULES 300 1.8 g (Active Comparator): EPADEL CAPSULES 300 0.9 g, orally, twice daily after breakfast and dinner for 12 weeks.
  Interventions: Drug: Icosapent (EPADEL CAPSULES 300)
- EPADEL CAPSULES 300 2.7 g (Active Comparator): EPADEL CAPSULES 300 0.9 g, orally, three-times daily after each meal for 12 weeks.
  Interventions: Drug: Icosapent (EPADEL CAPSULES 300)

INTERVENTIONS:
Drug: Icosapent (MND-2119) — Icosapent (MND-2119) capsules.
  Arms: MND-2119 2 g; MND-2119 4 g
Drug: Icosapent (EPADEL CAPSULES 300) — Icosapent (EPADEL CAPSULES 300) capsules.
  Arms: EPADEL CAPSULES 300 1.8 g; EPADEL CAPSULES 300 2.7 g

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of MND-2119 compared to EPADEL CAPSULES 300 in participants with hypertriglyceridemia.

DETAILED DESCRIPTION:
MND-2119 is a new formulation of Icosapent. This is a phase 3 study to evaluate the efficacy and safety of MND-2119 compared to EPADEL CAPSULES 300 in subjects with hypertriglyceridemia.

The study period is a total of 22 weeks and is comprised of 8 weeks run-in period, 12 weeks treatment period and 2 weeks follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Participants diagnosed with hypertriglyceridemia.
2. Participants with values of fasting triglyceride level are 150 mg/dL or higher and less than 500 mg/dL.

Exclusion Criteria:

1. Participants who have confirmed myocardial infarction and angina pectoris within 6 months.
2. Participants who have aortic aneurysm or has received aortic aneurysmectomy within 6 months.
3. Participants with, or with a history of, pancreatitis.
4. Participants who have a history or complication of a clinically significant hemorrhagic disease within 6 months.
5. Participants taking both anti-coagulants and anti-platelets.
6. Participants receiving dual antiplatelet therapy.
7. Participants taking direct oral anticoagulants.

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 580 (Actual)
Dates: Start 2018-10-27 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-06-29 (Actual)

PRIMARY OUTCOMES:
Percentage of change from baseline in serum triglyceride level at 12 weeks after the start of study drug administration | Baseline and 12 weeks

SECONDARY OUTCOMES:
Percentage of change from baseline in serum total cholesterol level at 12 weeks after the start of study drug administration | Baseline and 12 weeks
Percentage of change from baseline in serum low-density lipoprotein cholesterol (LDL-C) (direct method) level at 12 weeks after the start of study drug administration | Baseline and 12 weeks
Percentage of change from baseline in serum LDL-C (indirect method) level at 12 weeks after the start of study drug administration | Baseline and 12 weeks
Percentage of change from baseline in serum high-density lipoprotein cholesterol (HDL-C) level at 12 weeks after the start of study drug administration | Baseline and 12 weeks
Percentage of change from baseline in serum non HDL-C level at 12 weeks after the start of study drug administration | Baseline and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kohichi Hayashi, Study Director — Mochida Pharmaceutical Company, Ltd.
Locations (1):
- Mochida Investigational sites, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No